CLINICAL TRIAL: NCT06118359
Title: Development and Pilot Testing of an Intervention to Support Interhospital Transfer Decisions (SITe) Regarding Older Adults With Emergency General Surgery Diagnoses
Brief Title: Development and Pilot Testing the SITe Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator taking a new position.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-0838; 1R03AG078889-01 (NIH); Approval Date 6/23/2022 (Other: UW Madison); SMPH/SURGERY/TRAUMA (Other: UW Madison)
Record Dates: First submitted 2023-06-12; First posted 2023-11-07 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Emergency General Surgery
Keywords: Older adults; Communication; Health care provider; Interhospital transfer
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: The intervention will target UW Health accepting providers. Referring providers do not receive the intervention. Patients have waiver of informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SITe training for accepting providers (Experimental): UW Health (accepting) providers will participate in a training to learn how to utilize SITe intervention tools during EGS transfer calls.
  Interventions: Behavioral: Intervention to Support Interhospital Transfer Decisions (SITe)

INTERVENTIONS:
Behavioral: Intervention to Support Interhospital Transfer Decisions (SITe) — The SITe intervention and implementation toolkit was developed in Aim 1 through stakeholder activities. SITe, an intervention to support interhospital transfer decisions regarding older EGS patients, includes a checklist and script to be utilized by accepting providers during their conversations with referring providers. The investigators and stakeholders also developed a toolkit for implementation with resources to reduce barriers to and support facilitators of utilizing the tools. The toolkit includes: (1) the checklist and script; (2) methods to train accepting providers on the tools including a PowerPoint presentation and demonstration video; and (3) resources to familiarize other parties (transfer center nurses, referring providers, referring hospitals) with the SITe intervention.

SUMMARY:
Every year, nearly 240,000 patients age 60 and older are transferred between acute care hospitals for nontraumatic surgical emergencies, and these patients experience worse outcomes than patients admitted directly from an emergency department within a given hospital. Care coordination for older patients with emergency general surgery (EGS) diagnoses suffers because conversations between referring and accepting providers regarding decisions to transfer are ineffective, incomplete, and inefficient. To standardize a method to support transfer decisions that is tailored to older adults within extant transfer processes, the team will (1) engage key stakeholders to develop the intervention to Support Interhospital Transfer Decisions (SITe) for older EGS patients by adapting an existing intervention for interhospital handoffs and (2) assess the acceptability of the SITe intervention, test the feasibility of study procedures, and explore efficacy outcomes for evaluation in a future, larger clinical trial.

DETAILED DESCRIPTION:
Aim 2 of the protocol qualifies as a clinical trial. Aim 2 will assess the acceptability of the intervention to Support Interhospital Transfer Decisions (SITe), test the feasibility of study procedures, and explore efficacy outcomes for evaluation in a future, larger clinical trial. Modeling a similar and successful pilot, the investigators will conduct a pre (control)/post (intervention) study with 50 transfers in each arm. They will collect pre- and post-intervention data after each eligible transfer through (1) chart review and transfer center logs and (2) Qualtrics surveys of referring and accepting providers. The team will collect baseline (pre) and post-intervention measures of the potential to avoid transfers, efficiency of transfer communication and execution, provider emotional labor, and patient health outcomes. accepting providers will utilize the SITe intervention during calls discussing transfer decisions regarding older emergency general surgery patients. Transfer center nurses and referring providers will be informed of the SITe intervention tool.

The study was terminated early. The research team completed pre-intervention data collection and intervention training. No post-intervention data was collected. As of 3/21/2024, the UW-Madison IRB no longer considers training accepting surgeons on the intervention research.

ELIGIBILITY:
Inclusion Criteria:

* Patients (n=100): patients age 60 and older with an EGS diagnosis transferred from a referring ED or inpatient floor in Wisconsin to the UW ED or inpatient floor under care of UW surgeons
* Providers: all UW (accepting) surgeons and all referring providers who execute transfers of the 100 eligible patients. There will be no exclusions regarding referring providers' position (e.g., physician, mid-level provider), specialty (e.g., emergency medicine, internal medicine), or affiliation (e.g., UW or non-UW).

Exclusion Criteria:

* Providers who do not speak English
* Patients younger than 60 years
* Other interhospital transfers other than EGS transfers
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Ingraham, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the intervention training, 9 accepting surgeons were invited to be trained on the transfer tools; 3 accepting surgeons have accepted the invitation and were trained. Six accepting surgeons were invited but did not accept the invitation to complete the training. 25 unique providers took surveys, 3 accepting surgeons trained on the intervention were among them.
Pre-assignment Details: 60 calls met the initial screening criteria, 12 calls were excluded do to errors in screening, 48 transfer calls were eligible for 59 unique providers. Of those, 24 unique providers declined to take 28 surveys, and the team did not have contact information for 14 providers. Therefore 25 unique providers started the intervention.
Units Other Than Participants: Surveys
Groups:
- Referring Providers: Referring providers who called to discuss potential transfer of a patient (who was at least 60 years old with an emergency general surgery diagnosis) with an accepting provider
- Accepting Providers: Accepting providers who discussed potential transfer of a patient (who was at least 60 years old with an emergency general surgery diagnosis) with a referring provider
Period: Overall Study
Arm/Group | Referring Providers | Accepting Providers
Started (Unique providers identified to receive the survey.) | 13; 13 Surveys (47 unique referring providers asked to take 48 unique surveys.) | 12; 41 Surveys (12 unique accepting providers asked to take 48 unique surveys.)
Providers Enrolled in Intervention Training | 0; 0 Surveys (Survey units do not apply for Intervention Training) | 3; 0 Surveys (Survey units do not apply for Intervention Training)
Completed (Unique providers who completed the survey.) | 13; 13 Surveys | 12; 41 Surveys (All unique accepting providers took at least 1 survey, so there were 12 participants 'consented' by taking a survey. 41 completed surveys.)
Not Completed | 0; 0 Surveys | 0; 0 Surveys

BASELINE CHARACTERISTICS:
Population: 13 unique referring providers completed study survey, 12 unique accepting providers completed study surveys, and 3 accepting providers completed intervention training.
Groups:
- Total: Total of all reporting groups
Arm/Group | Referring Providers | Accepting Providers | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Full Range); unit: years] — Population: One accepting provider declined to provide age.
  years
    number analyzed (Participants) | 13 | 11 | 24
    (all) | 45.46 [31 to 68] | 45.4 [36 to 58] | 45.42 [31 to 68]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 10 | 5 | 15
  Woman | 2 | 7 | 9
  Non-binary | 0 | 0 | 0
  Prefer to self describe | 0 | 0 | 0
  Prefer not to say | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
Profession [Count of Participants; unit: Participants]
  Physician | 12 | 12 | 24
  Advanced Practice Provider (NP, PA) | 0 | 0 | 0
  Other | 1 | 0 | 1
Number of years practiced since training was finished [Mean (Full Range); unit: years] | 12.12 [0 to 32] | 10.2 [1 to 21] | 11.18 [0 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of the Intervention to Support Interhospital Transfer Decisions (SITe)
Description: The team will identify 50 study-eligible patient transfers post-intervention training.
  The team will ask the accepting provider and referring provider who executed the eligible transfer to rate the following statements on a Likert-scale (1=completely disagree to 5=completely agree):
  * This intervention meets my approval.
  * This intervention is appealing to me.
  * I like this intervention.
  * I welcome this intervention.
  Acceptability is defined as a minimum average score of 4 per item.
Time Frame: 3 months
Population: The study terminated early and the team mainly completed pre-intervention surveys and training activities. The study team did not complete post-intervention activities and analysis.
Groups:
- Accepting Providers Trained on SITe Tools: UW Health (accepting) providers will have been trained on the SITe intervention tools to use during EGS transfer calls. We will measure the acceptability of those tools by those providers.
Arm/Group | Accepting Providers Trained on SITe Tools
Number analyzed (Participants) | 0

2. Primary Outcome: Fidelity to the Intervention to Support Interhospital Transfer Decisions (SITe)
Description: The team will identify 50 study-eligible patient transfers post-intervention training. The team will measure missingness of the tool elements. Fidelity is defined as <15% missing patient information.
Time Frame: 3 months
Population: Study terminated early and these data were not collected.
Groups:
- Transfer Calls Taken by Accepting Providers Trained on SITe Tools: UW Health (accepting) providers will have been trained on the SITe intervention tools to use during EGS transfer calls. We will measure the fidelity to those tools by those providers.
Arm/Group | Transfer Calls Taken by Accepting Providers Trained on SITe Tools
Number analyzed (Participants) | 0

3. Primary Outcome: Feasibility of Study Procedures
Description: The team will measure the rate of survey completion for study-eligible patient transfers and examine rates of and reasons for missing outcome data.
Time Frame: pre-intervention at 3 months, post-intervention at 7 months
Population: Data was collected over 3 months prior to intervention, planned post-intervention data collection did not occur due to termination of the study.
Measure: Count of Units; unit: Surveys
Units Other Than Participants: Surveys
Arm/Group | Referring Providers | Accepting Providers
Number analyzed (Participants) | 13 | 12
Number analyzed (Surveys) | 34 | 48
Surveys
  Pre-Intervention Surveys | 13 | 41
  Post-Intervention Surveys: number analyzed (Participants) | 0 | 0
  Post-Intervention Surveys: number analyzed (Surveys) | 0 | 0
  Post-Intervention Surveys | 0 | 0

4. Primary Outcome: Potential to Avoid Transfer: Chart Review
Description: The team will evaluate the quality outcome: potential to avoid transfer. Through chart review, the team will look at number of transfers with no intervention and discharge to home within 72 hours.
Time Frame: 7 months
Population: Study terminated early and these data were not collected.
Groups:
- Calls Discussing Transfer - Before Intervention Training; Calls Discussing Transfer - After Intervention Training: Calls discussing transfer of patients who were at least 60 years old with an emergency general surgery diagnosis.
  UW Health (accepting) providers will participate in a training to learn how to utilize SITe intervention tools during EGS transfer calls.
  Intervention to Support Interhospital Transfer Decisions (SITe): The SITe intervention and implementation toolkit was developed in Aim 1 through stakeholder activities. SITe, an intervention to support interhospital transfer decisions regarding older EGS patients, includes a checklist and script to be utilized by accepting providers during their conversations with referring providers. The investigators and stakeholders also developed a toolkit for implementation with resources to reduce barriers to and support facilitators of utilizing the tools. The toolkit includes: (1) the checklist and script; (2) methods to train accepting providers on the tools including a PowerPoint presentation and demonstration video; and (3) resources to familiarize other parties (transfer center nurses, referring providers, referring hospitals) with the SITe intervention.
Arm/Group | Calls Discussing Transfer - Before Intervention Training | Calls Discussing Transfer - After Intervention Training
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Potential to Avoid Transfer- Second Related Question on Survey - Should Have Been Able
Description: The team will evaluate the quality outcome: potential to avoid transfer.
  Accepting Providers were asked: "I felt that the referring hospital should have been able to care for the patient." A similar question was not asked of Referring Providers
Time Frame: pre-intervention at 3 months, post-intervention at 7 months
Population: as for outcome 3
Measure: Number; unit: surveys
Units Other Than Participants: Surveys
Groups:
- Accepting Providers - Pre-Intervention: Accepting providers who discussed potential transfer of a patient (who was at least 60 years old with an emergency general surgery diagnosis) with a referring provider
Arm/Group | Accepting Providers - Pre-Intervention
Number analyzed (Participants) | 12
Number analyzed (Surveys) | 41
surveys
  Strongly agree | 4
  Agree | 12
  Neutral | 15
  Disagree | 8
  Strongly Disagree | 2

6. Primary Outcome: Efficiency of Transfer Communication
Description: Following the Relational Model of Organizational Change and through chart review and review of transfer center logs, the team will evaluate the efficiency of transfer communication. The team will review the number of calls required to complete the transfer and time required to complete transfer calls.
Time Frame: 7 months
Population: Study terminated early and these data were not collected.
Arm/Group | Calls Discussing Transfer - Before Intervention Training | Calls Discussing Transfer - After Intervention Training
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Efficiency of Transfer Execution
Description: The team will evaluate the efficiency of transfer execution. The team will review the time from initial call to patient arrival.
Time Frame: 7 months
Population: Study terminated early and these data were not collected.
Groups:
- Efficiency of Transfer Execution - Before Intervention Training; Efficiency of Transfer Execution - After Intervention Training: Time to transfer of patients who are at least 60 years old with an emergency general surgery diagnosis and transferred to UW Health.
  UW Health (accepting) providers will participate in a training to learn how to utilize SITe intervention tools during EGS transfer calls.
  Intervention to Support Interhospital Transfer Decisions (SITe): The SITe intervention and implementation toolkit was developed in Aim 1 through stakeholder activities. SITe, an intervention to support interhospital transfer decisions regarding older EGS patients, includes a checklist and script to be utilized by accepting providers during their conversations with referring providers. The investigators and stakeholders also developed a toolkit for implementation with resources to reduce barriers to and support facilitators of utilizing the tools. The toolkit includes: (1) the checklist and script; (2) methods to train accepting providers on the tools including a PowerPoint presentation and demonstration video; and (3) resources to familiarize other parties (transfer center nurses, referring providers, referring hospitals) with the SITe intervention.
Arm/Group | Efficiency of Transfer Execution - Before Intervention Training | Efficiency of Transfer Execution - After Intervention Training
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Emotional Labor - First Related Question on Survey - Respect
Description: Following the Relational Model of Organizational Change and specific Qualtrics questions, the team will evaluate the emotional labor of providers. The team will ask about providers' feelings about being listened to and supported when discussing patient care and difficult patient issues.
  Question for Referring Providers: I felt respected by the referring provider. Question for Accepting Providers: I felt respected by the UW surgeon.
Time Frame: pre-intervention at 3 months, post-intervention at 7 months
Population: as for outcome 3
Measure: Number; unit: surveys
Units Other Than Participants: Surveys
Groups:
- Referring Providers Pre-Intervention: Referring providers who called to discuss potential transfer of a patient (who was at least 60 years old with an emergency general surgery diagnosis) with an accepting provider
- Accepting Providers Pre-Intervention: Accepting providers who discussed potential transfer of a patient (who was at least 60 years old with an emergency general surgery diagnosis) with a referring provider
Arm/Group | Referring Providers Pre-Intervention | Accepting Providers Pre-Intervention
Number analyzed (Participants) | 13 | 12
Number analyzed (Surveys) | 13 | 41
surveys
  Strongly disagree | 0 | 0
  Disagree | 0 | 2
  Neutral | 2 | 5
  Agree | 5 | 24
  Strongly agree | 6 | 10

9. Primary Outcome: Patient Health Outcomes
Description: The team will evaluate patient health outcomes. The team will measure the number of admissions to the emergency department vs inpatient floor, the number of changes in level of patient care (general, intermediate, intensive) within 24 hours of arrival, and the number of adverse events (inpatient mortality, morbidity, extended length of stay.)
Time Frame: 7 months
Population: Study terminated early and these data were not collected.
Groups:
- Patient Health Outcomes - Before Intervention Training; Patient Health Outcomes - After Intervention Training: UW Health (accepting) providers will participate in a training to learn how to utilize SITe intervention tools during EGS transfer calls.
  Intervention to Support Interhospital Transfer Decisions (SITe): The SITe intervention and implementation toolkit was developed in Aim 1 through stakeholder activities. SITe, an intervention to support interhospital transfer decisions regarding older EGS patients, includes a checklist and script to be utilized by accepting providers during their conversations with referring providers. The investigators and stakeholders also developed a toolkit for implementation with resources to reduce barriers to and support facilitators of utilizing the tools. The toolkit includes: (1) the checklist and script; (2) methods to train accepting providers on the tools including a PowerPoint presentation and demonstration video; and (3) resources to familiarize other parties (transfer center nurses, referring providers, referring hospitals) with the SITe intervention.
Arm/Group | Patient Health Outcomes - Before Intervention Training | Patient Health Outcomes - After Intervention Training
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Emotional Labor - Second Related Question on Survey - Listening
Description: Following the Relational Model of Organizational Change and specific Qualtrics questions, the team will evaluate the emotional labor of providers. The team will ask about providers' feelings about being listened to and supported when discussing patient care and difficult patient issues.
  Question for Referring Providers: The UW Surgeon listened to my concerns about the patient.
  A similar question was not asked of Accepting Providers
Time Frame: pre-intervention at 3 months, post-intervention at 7 months
Population: as for outcome 3
Measure: Number; unit: surveys
Units Other Than Participants: Surveys
Arm/Group | Referring Providers Pre-Intervention
Number analyzed (Participants) | 13
Number analyzed (Surveys) | 13
surveys
  Strongly disagree | 0
  Disagree | 1
  Neutral | 0
  Agree | 5
  Strongly agree | 7

11. Primary Outcome: Emotional Labor - Third Related Question on Survey - Understanding
Description: Following the Relational Model of Organizational Change and specific Qualtrics questions, the team will evaluate the emotional labor of providers. The team will ask about providers' feelings about being listened to and supported when discussing patient care and difficult patient issues.
  Question for Referring Providers: I felt that the UW Surgeon understood my reason for transfer.
  A similar question was not asked of Accepting Providers
Time Frame: pre-intervention at 3 months, post-intervention at 7 months
Population: as for outcome 3
Measure: Number; unit: surveys
Units Other Than Participants: Surveys
Arm/Group | Referring Providers Pre-Intervention
Number analyzed (Participants) | 13
Number analyzed (Surveys) | 13
surveys
  Strongly disagree | 0
  Disagree | 1
  Neutral | 0
  Agree | 5
  Strongly agree | 7

12. Primary Outcome: Emotional Labor - Fourth Related Question on Survey - Doubt
Description: Following the Relational Model of Organizational Change and specific Qualtrics questions, the team will evaluate the emotional labor of providers. The team will ask about providers' feelings about being listened to and supported when discussing patient care and difficult patient issues.
  Question for Referring Providers: I felt that the UW Surgeon doubted whether the transfer was necessary.
  A similar question was not asked of Accepting Providers
Time Frame: pre-intervention at 3 months, post-intervention at 7 months
Population: as for outcome 3
Measure: Number; unit: surveys
Units Other Than Participants: Surveys
Arm/Group | Referring Providers Pre-Intervention
Number analyzed (Participants) | 13
Number analyzed (Surveys) | 13
surveys
  Strongly disagree | 8
  Disagree | 4
  Neutral | 0
  Agree | 0
  Strongly agree | 1

13. Primary Outcome: Potential to Avoid Transfer- First Related Question on Survey - Justifiable
Description: The team will evaluate the quality outcome: potential to avoid transfer.
  Accepting Providers were asked: "I felt that the reason for transfer was justifiable." A similar question was not asked of Referring Providers
Time Frame: pre-intervention at 3 months, post-intervention at 7 months
Population: as for outcome 3
Measure: Number; unit: surveys
Units Other Than Participants: Surveys
Arm/Group | Accepting Providers Pre-Intervention
Number analyzed (Participants) | 12
Number analyzed (Surveys) | 41
surveys
  Strongly Disagree | 3
  Disagree | 4
  Neutral | 13
  Agree | 13
  Strongly agree | 8

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected for this study
Description: Adverse event data were not collected for this study
Arm/Group | SITe Training for Accepting Providers
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Although the study team did complete pre-intervention activities and implemented the intervention (training of accepting providers), most outcome data were not collected because the study ended prematurely. The team was not able to collect post-intervention data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT06118359/Prot_000.pdf
  • Informed Consent Form (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT06118359/ICF_001.pdf